CLINICAL TRIAL: NCT04387929
Title: Observational Cohort Study for the Detection of Anti-COVID-19 Antibody Levels in an Hospital Population
Brief Title: Detection of Anti-COVID-19 Antibody Levels in an Hospital Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1374 IgG COVID-19 HUMANITAS
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; Antibody titer; Serological tests; Hospital personnel
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IgG negative: No intervantion. Only antibody mesurment from blood sample
  Interventions: Diagnostic Test: Detection of anti-COVID-19 antibody level
- IgG positive, viral load negative: No intervantion. Only antibody mesurment from blood sample and viral load from nasopharyngeal swabs
  Interventions: Diagnostic Test: Detection of anti-COVID-19 antibody level
- IgG positive, viral load positive: No intervantion. Only antibody mesurment from blood sample and viral load from nasopharyngeal swabs
  Interventions: Diagnostic Test: Detection of anti-COVID-19 antibody level

INTERVENTIONS:
Diagnostic Test: Detection of anti-COVID-19 antibody level — Detection of anti-COVID-19 antibody level form blood samples. If positive, viral load will be measured by RT-PCR of nasopharyngeal swab.

SUMMARY:
COVID-19 (SARS-CoV-2) infection in health professionals represent a significant criticality both for the risk of spreading the disease and for the organizational aspects that follow. The objective of the study is to evaluate the spread of COVID-19 virus within the hospital population of Humanitas through the monitoring of the levels of IgG antibodies. Moreover, viral load will be measured by RT-PCR in the subgroup positive to IgG antibodies.

DETAILED DESCRIPTION:
The Coronavirus identified in Wuhan, China, for the first time in late 2019 is a new viral strain that has never previously been identified in humans. It has been called SARS-CoV-2 and the respiratory disease that causes COVID-19. SARS-CoV-2 infection in health professionals has represented and continues to represent a significant criticality both for the risk of spreading the disease and for the organizational aspects that follow.

Currently the gold standard for the non-invasive diagnosis of COVID-19 is the detection of the viral genome by RT-PCR. However, despite the high specificity, this technique has a low sensitivity and can produce false negative samples. Furthermore, detection of the viral genome is indicative of active infection and fails to identify subjects previously exposed to the virus who have passed the infection asymptomatically. Serological tests can detect the presence of anti-SARS-CoV-2 antibodies in blood or serum samples and, depending on the type of antibody detected, identify the subjects in the active phase of the infection and after the resolution of the infection, the whose diagnosis was not made by performing a swab.

We will evaluate the actual spread of the SARS-CoV-2 virus within the hospital personnel of Humanitas through the monitoring of the levels of IgG antibodies. Moreover, viral load will be measured by RT-PCR of nasopharyngeal swabs in the subgroup positive to IgG antibodies. Secondary endpoints are: visualize the trend of the antibody value at 3, 6 and 12 months; correlation between the antibody titer in test positive subjects and the viral load of the nasopharyngeal swab; identification of predictive variables of susceptibility to viral SARS-CoV2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* work for the Humanitas Group (Rozzano / San Pio X, Humanitas Gavazzeni, Humanitas Mater Domini, Humanitas University, Humanitas Medical Care)
* Work activity in the Humanitas Group for at least 3 months among which, for example:

Healthcare Staff (Doctors, Nurses, OSS) Technical Staff (Biologists, Radiology Technicians, Laboratory Technicians, etc.) PARC staff and Staff Staff Research Internship students of Hunimed Contract staff (e.g. transport and sanitation services)

* Signature of informed consent
* Compilation of the anamnestic questionnaire

Exclusion Criteria:

* Subjects absent for any reason during the study period

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Personnel of Humanitas Group including:
  Healthcare Staff (Doctors, Nurses, OSS) Technical Staff (Biologists, Radiology Technicians, Laboratory Technicians, etc.) PARC staff and Staff Staff Research Internship students of Hunimed Contract staff (e.g. transport and sanitation services)
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 levels of IgG antibodies | 1 year
  Measurement of the temporal trend of the antibody value of anti-SARS-CoV-2 neutralizing IgG.

SECONDARY OUTCOMES:
SARS-CoV-2 viral load in nasopharyngeal swab of IgG positive subjects | 1 year
  Measurement of the viral load of the nasopharyngeal swab in antibody test positive subjects and the correlation between the antibody titer and virus positivity or negativity.
Epidemiology correlations | 1 year
  The association between the antibody value and potential protective or risk factors of the subject participating in the study such as age, clinical history, vaccination history, workplace, professional category, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Rozzano/San Pio X, Rozzano, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levi R, Azzolini E, Pozzi C, Ubaldi L, Lagioia M, Mantovani A, Rescigno M. One dose of SARS-CoV-2 vaccine exponentially increases antibodies in individuals who have recovered from symptomatic COVID-19. J Clin Invest. 2021 Jun 15;131(12):e149154. doi: 10.1172/JCI149154. PMID 33956667